CLINICAL TRIAL: NCT00673179
Title: Outpatient Chemotherapy in Pediatric Osteosarcoma: Doxorubicin With Cisplatin, High-Dose Methotrexate, and Additional Risk-Adapted Outpatient Chemotherapy
Brief Title: Doxorubicin With Cisplatin, High-Dose Methotrexate, and Additional Risk-Adapted Outpatient Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0404
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Osteosarcoma
Keywords: Doxorubicin; AD; Hydroxydaunomycin hydrochloride; Cisplatin; Paraplatin®; Methotrexate; Ifosfamide; Osteosarcoma; Sargramostim; Leukine™; Leucovorin; Gemcitabine; Gemzar; Gemcitabine Hydrochloride; GM-CSF; Questionnaire; Survey
MeSH Terms: conditions — Osteosarcoma | interventions — Doxorubicin; Cisplatin; Carboplatin; Methotrexate; Leucovorin; Dexrazoxane; Ifosfamide; Surveys and Questionnaires; Gemcitabine; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Surgical Procedures, Operative; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Chemotherapy (Experimental): Pre-Surgery, Regimen 1: Doxorubicin intravenous (IV) 90 mg daily, Cisplatin 60 mg/m^2/day for 2 days, Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Surgery; Post-Surgery, Regimen 1: Methotrexate 12 gm/m^2, Doxorubicin IV 90 mg, Cisplatin 60 mg/ m^2 twice daily, Leucovorin Rescue.
  Interventions: Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate; Drug: Leucovorin; Behavioral: Questionnaire; Procedure: Surgery
- Additional Risk-Adapted Outpatient Chemotherapy (Experimental): Pre-Surgery, Regimen 2: Dexrazoxane 900 mg/m^2 intravenous (IV) then Doxorubicin IV 90 mg daily, Cisplatin 120 mg/m^2 (intra-arterial); Surgery; Post-Surgery, Regimen 2: Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Ifosfamide 2.8 grams m^2/day and Mesna 2.8 gm/m^2/day continuous IV over 6 days; Lung-Directed Chemotherapy, Regimen 2: Gemcitabine, Sargramostim Inhaled aerosol (5 mcg/kg, maximum dose 300 mcg).
  Interventions: Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate; Drug: Leucovorin; Drug: Dexrazoxane; Drug: Ifosfamide; Behavioral: Questionnaire; Drug: Gemcitabine; Drug: Sargramostim; Procedure: Surgery; Drug: Mesna

INTERVENTIONS:
Drug: Doxorubicin — Pre-Surgery, Regimen 1: IV Over 15 Minutes on Day 1 of Weeks 1 and 6; Post-Surgery, Regimen 1: IV on Day 1 of Weeks 16, 21, and 26; Pre-Surgery, Regimen 2: IV over 15 Minutes on Day 1 of Weeks 1, 4, and 7. Dose 90 mg/m^2.
  Other Names: AD; Hydroxydaunomycin hydrochloride
Drug: Cisplatin — Pre-Surgery, Regimen 1: IV Over 48 Hours, on Days 1 and 2 of Weeks 1 and 6; Post-Surgery, Regimen 1: IV Over 48 Hours, on Days 1 and 2 of Weeks 16, 21, and 26. Pre-Surgery, Regimen 2: Infusion through an artery over 4 hours on Day 1 of Weeks 1, 4, and 7. Dose 60 mg/m^2/day for 2 days continuous infusion.
  Other Names: Paraplatin®
Drug: Methotrexate — Pre-Surgery, Regimen 1: IV Over 4 Hours on Day 1 of Weeks 4, 5, 9, and 10; Post-Surgery, Regimen 1: IV Over 4 Hours on Day 1 of Weeks 14, 15, 19, 20, 24, 25, 29, and 30; Post-Surgery, Regimen 2: IV Over 4 Hours on Day 1 of Weeks 14, 15, 20, 21, 26, 27, 32, 33, 38, and 39. Dose 12 gm/m^2, max 20 gm over 4 hours.
Drug: Leucovorin — Pre- and Post-Surgery, Regimen 1: IV Over 5 minutes on the day after each methotrexate dose and then by mouth every 6 hours; Post-Surgery, Regimen 2: IV Over 5 minutes on the day after each methotrexate dose and then by mouth every 6 hours. Dose 10 mg IV, with 10 mg orally every 6 hours.
Drug: Dexrazoxane — Dose 900 mg/m^2 IV Push with doxorubicin. Pre-Surgery, Regimen 2: IV Over 15 minutes on Day 1 of Weeks 1, 4, and 7.
  Other Names: Zinecard
  Arms: Additional Risk-Adapted Outpatient Chemotherapy
Drug: Ifosfamide — Post-Surgery, Regimen 2: IV continuously over 5 days each time, on Weeks 16, 22, 28, and 34. Dose 2.8 gm/m^2. Dose 2.8 grams m^2/day.
  Other Names: Ifex
  Arms: Additional Risk-Adapted Outpatient Chemotherapy
Behavioral: Questionnaire — Questionnaires to be completed on 5 different days during the study.
  Other Names: Survey
Drug: Gemcitabine — IV over 1 hour, every other week.
  Other Names: Gemzar; Gemcitabine Hydrochloride
  Arms: Additional Risk-Adapted Outpatient Chemotherapy
Drug: Sargramostim — Inhaled aerosol (5 mcg/kg, maximum dose 300 mcg) twice a day for 7 days on, 7 days off, beginning the day receive gemcitabine.
  Other Names: GM-CSF; Leukine™
  Arms: Additional Risk-Adapted Outpatient Chemotherapy
Procedure: Surgery — Planned limb salvage surgery after 3 courses of doxorubicin + cisplatin (IV) and High-dose methotrexate - at approximately week 12.
Drug: Mesna — IV continuously over 6 days each time, on Weeks 16, 22, 28, and 34. Dose 2.8 gm/m^2/day.
  Other Names: Mesnex
  Arms: Additional Risk-Adapted Outpatient Chemotherapy

SUMMARY:
The goal of this clinical research study is to learn if giving certain combinations of chemotherapy drugs before and after surgery, mostly in the outpatient clinic instead of in the hospital, can result in fewer hospital stays during treatment for osteosarcoma. The drugs and schedules will vary depending on the status of the cancer and its level of risk for spreading, but they will include combinations of doxorubicin (non-liposomal), cisplatin, methotrexate, and ifosfamide, as described below.

DETAILED DESCRIPTION:
The Study Drugs:

The standard treatment combination used to treat patients with osteosarcoma is doxorubicin, cisplatin, and methotrexate with or without ifosfamide. When this treatment combination is given in the hospital, it can require around 18-22 hospital stays. Somewhat recently, chemotherapy for osteosarcoma has become possible to give in the outpatient clinic. Researchers want to learn if giving 4 certain drugs (the combination of doxorubicin, cisplatin, and methotrexate with or without ifosfamide) in the outpatient setting to eligible patients will help to decrease the number of hospital stays.

During this study, all study participants whose tumor(s) can be taken out with surgery will be offered routine surgery to remove the tumor(s). After surgery, if the doctor believes the tumor(s) have responded well enough, the standard treatment combination is again doxorubicin, cisplatin, and methotrexate. If the tumor(s) have not responded well enough, however, the standard treatment combination is methotrexate and ifosfamide.

In this study, participants are considered at "higher risk" for the tumor(s) spreading to the lungs in the following cases: if the participant's tumor(s) are large at the time of joining this study, if the cancer has spread to other organs, and/or if standard chemotherapy in this study has not killed enough tumor cells.

The following drugs are used in this study:

* Doxorubicin is designed to stop the growth of cancer cells, which may cause the cells to die.
* Cisplatin has an atom at its center that contains a type of metal called platinum. The platinum is supposed to poison the cancer cells.
* Methotrexate is designed to disrupt cells (including cancer cells) from making and repairing DNA and "copying" themselves.
* Ifosfamide is designed to stop the growth of cancer cells, which may cause the cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 groups based on the likelihood that the surgery will be able to control the disease in the arm or leg that has the bone tumor(s).

Group 1 includes participants who are considered to have a "standard" chance that surgery will be able to control the disease in the arm or leg, participants who will have an amputation, or participants with cancer in areas other than in an arm or leg at the time of diagnosis.

Group 2 includes participants who are considered to have a "higher" chance that the tumor(s) will be left behind after having surgery that the doctor considers as "incomplete" to control the disease.

Central Venous Line:

For drugs to be given by vein, your study doctor will likely recommend that you have a central venous line (CVL) placed. A central venous line is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Pre-Surgery Chemotherapy for Group 1:

Before surgery, Group 1 participants will receive doxorubicin, cisplatin, and methotrexate followed by leucovorin. Leucovorin is given to help prevent and/or treat the side effects that methotrexate may cause. Dexrazoxane is used to decrease the risk of side effects to the heart that doxorubicin may cause. These drugs will be given in an outpatient clinic (without requiring hospitalization), if possible.

Doxorubicin will be given by vein over 15 minutes, after dexrazoxane by vein over 15 minutes, on Day 1 of Weeks 1 and 6.

Cisplatin will be given as a continuous infusion by vein over 48 hours, on Days 1 and 2 of Weeks 1 and 6.

Methotrexate will be given by vein, over 4 hours, on Day 1 of Weeks 4, 5, 9, and 10. If you have difficulty recovering from the effects of the methotrexate therapy, you may only receive methotrexate twice before surgery, instead of 4 times.

Leucovorin will be given by vein, over 5 minutes, on the day after each methotrexate dose and then by mouth every 6 hours after that, until the study doctor believes that the methotrexate level in the blood is low. The methotrexate level in the blood will be checked using a blood test (less than 2 teaspoons each time). This test will be performed once a day after each methotrexate infusion, until the methotrexate blood level is low and it is considered safe to stop the leucovorin.

Pre-Surgery Chemotherapy for Group 2:

Before surgery, Group 2 participants will receive dexrazoxane, doxorubicin, and cisplatin.

On Day 1 of Weeks 1, 4, and 7, dexrazoxane will be given by vein over 15 minutes, followed by doxorubicin given by vein over 15 minutes and then cisplatin through an artery over 4 hours. Infusion through an artery requires a hospital stay of 2-4 days.

Surgery:

For all eligible study participants, the surgery to remove the tumor(s) will be performed on either Week 11 or 12. The surgery will be explained to you in detail, and you will be asked to sign a separate consent form for it that will describe its risks.

Before surgery, you will have routine visits with the surgeon. You will have several routine scans performed to help plan the surgery.

Chemotherapy Regimens after Surgery:

After the surgery (on or around Week 14), you will receive additional "post-surgery" chemotherapy.

After surgery, if you were originally in Group 1, and if the doctor believes the tumor(s) have responded well enough (specifically, if 90% or more of the tumor cells are dead when checked under the microscope), you will receive additional chemotherapy that is similar to what you received before surgery. This is described below as Regimen A. If the doctor does not believe the tumor(s) have responded well enough (if less than 90% of the tumor cells are dead when checked under the microscope), however, you will be assigned to Regimen B.

All participants who started in Group 2 will be assigned to Regimen B.

Radiation and Chemotherapy for Patients Ineligible for Routine Surgery:

A small number of participants on this study may need to have radiation therapy to help control the disease, as part of their routine care. This would only be done if the tumor(s) cannot be completely taken out with surgery, or if amputation is necessary but refused by the participant. If needed, and depending on where the tumor(s) are located, your doctor may decide that radiation is needed. All participants needing radiation or having surgery that the doctor considers as "incomplete" to control the disease are considered "higher risk" and will receive Regimen B therapy during and after radiation. (Radiation will usually begin during Weeks 12-14, but it could be anytime during ifosfamide therapy.) The radiation therapy will be explained to you in detail, and you will be asked to sign a separate consent form for it that will describe its risks.

Post-Surgery Chemotherapy for Regimen A:

Regimen A includes the following treatments:

* Methotrexate will be given over 4 hours on Day 1 of Weeks 14, 15, 19, 20, 24, 25, 29, and 30.
* Doxorubicin will be given on Day 1 of Weeks 16, 21, and 26.
* Cisplatin will be given as a continuous infusion by vein over 48 hours, on Days 1 and 2 of Weeks 16, 21, and 26.
* Leucovorin will be given by vein, over 5 minutes, on the day after each methotrexate dose and then by mouth every 6 hours after that, until the study doctor believes that the methotrexate level in the blood is low. The methotrexate level in the blood will be checked using a blood test (less than 2 teaspoons each time). This test will be performed once a day after each methotrexate infusion, until the methotrexate blood level is low and it is considered safe to stop the leucovorin.

Post-Surgery Chemotherapy for Regimen B:

Regimen B includes the following treatments:

* Methotrexate will be given over 4 hours on Day 1 of Weeks 14, 15, 20, 21, 26, 27, 32, 33, 38, and 39.
* Leucovorin will be given by vein, over 5 minutes, on the day after each methotrexate dose and then by mouth every 6 hours after that, until the study doctor believes that the methotrexate level in the blood is low. The methotrexate level in the blood will be checked using a blood test (less than 2 teaspoons each time). This test will be performed once a day after each methotrexate infusion, until the methotrexate blood level is low and it is considered safe to stop the leucovorin.
* Ifosfamide will be given by vein, continuously over 5 days each time, on Weeks 16, 22, 28, and 34.
* Mesna will be given by vein, continuously over 6 days each time, on Weeks 16, 22, 28, and 34. Mesna is used to decrease the risk of bleeding in the bladder and kidneys while ifosfamide is taken.

Study Tests:

After Week 5 of treatment, and then again before surgery, you will have the following tests performed:

* Your medical history will be reviewed.
* You will have a physical exam.
* Blood (about 2-3 teaspoons each time) will be collected for routine tests and tests of your kidney and liver function. The routine blood tests may be repeated more often during the weeks you are receiving any of the study drugs.

If you are receiving cisplatin, you may have a hearing test performed before each dose of this drug.

You will have an ECHO performed before your fourth dose of doxorubicin on Week 14, and possibly more often if necessary.

Questionnaires:

You will be asked to complete 5 brief questionnaires on 5 different days during this study. The questionnaires ask about the health-related quality of your life, and include questions about how you have felt, physically and emotionally, during cancer treatment. The questionnaires also ask how you and your family have adapted to your having cancer treatments, and what effects the medicines may have had on whether you have felt healthy or sick.

These questionnaires will be completed at Week 1, at about Week 7 (before surgery or radiation), sometime during Weeks 20-22, at the end-of-treatment visit (either the end-of-Regimen-A visit, the end-of-Regimen-B visit, or the end-of-treatment visit), and 1 year after your first diagnosis of cancer. It should take you about 15-20 minutes to fill out the questionnaires each time.

External Care:

If the study doctor allows and you agree, some of the blood tests in this study may be performed outside of M. D. Anderson. The study doctor will discuss this option with you, if applicable.

Length of Study Participation:

If the disease gets worse or intolerable side effects occur, you will be taken off study.

End-of-Regimen-A Visit, End-of-Regimen-B Visit, or End-of-Treatment Visit:

If you complete Regimen A or B as planned or you leave the study early for any reason, the following procedures will be performed:

* You will have a physical exam.
* Urine and blood (about 2-3 teaspoons) will be drawn for routine tests and tests of your kidney and liver function.
* You will have an ECHO, x-rays of the disease area and the chest, CT scans of the chest, and a bone scan.
* You will also have whole-body scans and a hearing test.

Follow-Up Visits:

After the end-of-Regimen-A visit, the end-of-Regimen-B visit, or the end-of-treatment visit, you will be asked to return for follow-up visits. At these visits, the following procedures will be performed:

* CT scans of the chest will be performed every 3 months for the first year after your chemotherapy ends, every 4 months for the 2nd year, every 6 months for the 3rd year, and once a year for the next 2 years.
* You will have a bone scan every year for 5 years.

This is an investigational study. All of the drugs used in this study are commercially available and commonly used in osteosarcoma. This study is designed to look at the drugs' use in the outpatient setting, which is considered research.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed high-grade osteosarcoma. Patients with unresectable or metastatic disease ARE eligible.
2. Age 5-40 years old on date of diagnostic biopsy.
3. Adequate organ function: creatinine 1.6 or lower, bilirubin <2, Hemoglobin 8 gm/dL or greater, Absolute neutrophil count (ANC) 1000 or more, platelets 100,000 or more. Cardiac ejection fraction (EF) 50% or better, hearing threshold 40 dB at 4000 Hz or better.
4. Signed informed consent.
5. Negative pregnancy test in females of child bearing potential, and if sexually active, willingness to use effective contraception during chemotherapy.

Exclusion Criteria:

1. Diagnosis other than osteosarcoma.
2. Pregnant or lactating females, or unwilling to use effective contraception during chemotherapy

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Anderson, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 05, 2008 to November 24, 2010. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Early study termination with low accrual.
Groups:
- Outpatient Chemotherapy: Pre-Surgery, Group 1: Doxorubicin intravenous (IV) 90 mg daily, Cisplatin 60 mg/m^2/day for 2 days, Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Surgery; Post-Surgery, Regimen A: Methotrexate 12 gm/m^2, Doxorubicin IV 90 mg, Cisplatin 60 mg/ m^2 twice daily, Leucovorin Rescue or Regimen B: Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Ifosfamide 2.8 grams m^2/day and Mesna 2.8 gm/m^2/day continuous IV over 6 days; Lung-Directed Chemotherapy, Regimen B: Gemcitabine, Sargramostim Inhaled aerosol (5 mcg/kg, maximum dose 300 mcg).
- Additional Risk-Adapted Outpatient Chemotherapy: Pre-Surgery, Group 2: Dexrazoxane 900 mg/m^2 intravenous (IV) then Doxorubicin IV 90 mg daily, Cisplatin 120 mg/m^2 (intra-arterial); Surgery; Post-Surgery, all Group 2 assigned to Regimen B: Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Ifosfamide 2.8 grams m^2/day and Mesna 2.8 gm/m^2/day continuous IV over 6 days; Lung-Directed Chemotherapy, Regimen 2: Gemcitabine, Sargramostim Inhaled aerosol (5 mcg/kg, maximum dose 300 mcg).
Period: Overall Study
Arm/Group | Outpatient Chemotherapy | Additional Risk-Adapted Outpatient Chemotherapy
Started | 7 | 0
Completed | 4 | 0
Not Completed | 3 | 0
Not completed — Toxicity/Complications | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Chemotherapy | Additional Risk-Adapted Outpatient Chemotherapy | Total
Number analyzed (Participants) | 7 | 0 | 7
Age, Continuous [Median (Full Range); unit: years] | 14 [11 to 18] |  | 14 [11 to 18]
Gender [Number; unit: participants]
  Female | 3 |  | 3
  Male | 4 |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success (6 or Fewer Hospitalizations During Front-line Chemotherapy)
Description: Treatment success defined as a patient having 6 or fewer hospitalizations during front-line chemotherapy.
Time Frame: Baseline to 5 Years
Population: Study terminated early without analysis.
Arm/Group | Outpatient Chemotherapy | Additional Risk-Adapted Outpatient Chemotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life (Ped QL) Assessment
Time Frame: Peds QL measures at week 0 (during first chemo cycle), week 6, week 20, at end of therapy, and at 3 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event reporting up to 39 weeks of varying treatment, with overall study 2 years, 2 months.
Description: Expected toxicities for these varieties of osteosarcoma chemotherapy.
Groups:
- Additional Risk-Adapted Outpatient Chemotherapy: Pre-Surgery, Group 2: Dexrazoxane 900 mg/m^2 intravenous (IV) then Doxorubicin IV 90 mg daily, Cisplatin 120 mg/m^2 (intra-arterial); Surgery; Post-Surgery, all Group 2 assigned to Regimen B: Methotrexate 12 gm/m^2, Leucovorin Rescue 10 mg IV, with 10 mg orally every 6 hours; Ifosfamide 2.8 grams m^2/day and Mesna 2.8 gm/m^2/day continuous IV over 6 days
Arm/Group | Outpatient Chemotherapy | Additional Risk-Adapted Outpatient Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/0
Other Adverse Events (participants affected / at risk) | 1/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Outpatient Chemotherapy (N=7) | Additional Risk-Adapted Outpatient Chemotherapy (N=0)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Outpatient Chemotherapy (N=7) | Additional Risk-Adapted Outpatient Chemotherapy (N=0)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 2

LIMITATIONS AND CAVEATS:
Study could not meet accrual goal due to logistical considerations, terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No